CLINICAL TRIAL: NCT01688882
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group Study Evaluating the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of QGE031 in the Treatment of Patients With Bullous Pemphigoid With Disease Refractory to Oral Steroid Treatment
Brief Title: Safety, Efficacy and PK/PD of QGE031 vs. Placebo in Patients With Active Bullous Pemphigoid Despite Oral Steroid Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was stopped after Part 1 completed and was terminated because the predefined criteria of efficacy was not reached ( >50% better then placebo)
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQGE031X2202
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: Bullous Pemphigoid
Keywords: bullous pemphigoid; QGE031
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — ligelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- QGE031 (Experimental): QGE031 240 mg Q2W s.c.
  Interventions: Drug: QGE031
- Placebo (Placebo Comparator): Placebo to Match Q2W s.c.
  Interventions: Drug: Placebo
- Open Label QGE031 (Experimental): Open Label QGE031 Q2W s.c.
  Interventions: Drug: QGE031

INTERVENTIONS:
Drug: QGE031 — QGE031 will be evaluated at various dose levels and regimens, based on the impact on disease of the next highest dose level and regimen.
  Arms: Open Label QGE031; QGE031
Drug: Placebo — Placebo will be used to control for normal variability in disease severity.
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of QGE031 versus placebo in patients with bullous pemphigoid. Efficacy will be assessed as a reduction of disease activity. How QGE031 is broken down by the body and the impact it has on different blood and tissue markers will also be explored.

DETAILED DESCRIPTION:
This study was planned to be divided into 2 distinct parts. Part 1 was a multicenter, randomized, placebo-controlled study evaluating the efficacy, safety, PK and PD of multiple, subcutaneous doses of QGE031 in the treatment of patients with BP with disease refractory to oral steroid treatment. Patients were treated with QGE031 or placebo in a 2:1 ratio.

Part 2 of this study was planned to be a multi-center, open label, dose range finding study evaluating the efficacy, safety, PK and PD of multiple, subcutaneous doses of QGE031 in the treatment of patients with BP with disease refractory to oral steroid treatment.

This study was stopped after Part 1 completed and was terminated because the predefined criteria of efficacy was not reached ( >50% better then placebo)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bullous pemphigoid
* Stable dose of prednisone at or above 10mg per day but no greater than 1 mg/kg/day
* Weigh between 40-120kg
* total IgE level up to 5000 IU/mL

Exclusion Criteria:

* Use of rituximab within 1 year

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (2):
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Durham, North Carolina
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Rouen, Cedex, France
- Germany (3):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Marburg
- Novartis Investigative Site, Shinjuku-ku, Tokyo, Japan
- Novartis Investigative Site, Taipei, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QGE031 | Placebo
Started | 13 | 7 (4 patients who completed 12 weeks of placebo changed to open-label QGE031 treatment.)
Safety Follow-up | 11 | 5
Completed | 10 | 6 (The one patient that discontinued was already switched to open-label QGE031 treatment.)
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 1
Not completed — Administrative problems | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QGE031 | Placebo | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (14.85) | 67.9 (14.60) | 65.2 (14.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 10 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Had a Clinical Global Assessment of Change (CGA-C) Responder Rate by Week 12
Description: Clinical Global Assessment of Change (CGA-C) responder rate was the responder rate at 12 weeks based on the CGA-C in bullous pemphigoid (BP).
  A patient with a CGA-C score of 3 or 4 indicating 'at least marked improvement from baseline' at 12 weeks was considered a responder. The CGA-C is an investigator assessment of change from baseline and is scored as follows: -4 = Very marked worsening (100% worsening); -3 = Marked worsening (67-99% worsening); -2 = Moderate worsening (34-66% worsening); -1 = Slight worsening (1-33% worsening); 1= Slight improvement (1-33% improvement); 2 = Moderate improvement (34-66% improvement); 3 = Marked improvement (67-99% improvement); 4 = Complete clearance (100% improvement)
Time Frame: 12 weeks
Population: Pharmacodynamics (PD) analysis set included all randomized patients.
Measure: Number; unit: number of participants
Arm/Group | QGE031 | Placebo
Number analyzed (Participants) | 13 | 7
number of participants | 8 | 2

2. Secondary Outcome: Response Based on Clinical Global Assessment of Change CGA-C Score at 6 Weeks
Description: Clinical Global Assessment of Change (CGA-C) responder rate was the responder rate at 6 weeks based on the CGA-C score in bullous pemphigoid (BP).
  A patient with a CGA-C score of 3 or 4 indicating marked improvement from baseline at 6 weeks was considered a responder. The CGA-C is an investigator assessment of change from baseline and is scored as follows: -4 = Very marked worsening (100% worsening); -3 = Marked worsening (67-99% worsening); -2 = Moderate worsening (34-66% worsening); -1 = Slight worsening (1-33% worsening); 1= Slight improvement (1-33% improvement); 2 = Moderate improvement (34-66% improvement); 3 = Marked improvement (67-99% improvement); 4 = Complete clearance (100% improvement)
Time Frame: 6 weeks
Population: Pharmacodynamics (PD) analysis set included all randomized patients.
Measure: Number; unit: number of participants
Arm/Group | QGE031 | Placebo
Number analyzed (Participants) | 13 | 7
number of participants | 8 | 2

3. Secondary Outcome: Number of Patients Investigator Global Assessment Score Over 12 Weeks
Description: Investigator's Global Assessment (IGA) - (scale of 0 to 4, where 0=clear, 1=almost clear, 2=mild, 3=moderate and 4=severe)
Time Frame: Baseline (week 0), week 6 and week 12
Population: Pharmacodynamics (PD) analysis set included all randomized patients.
Measure: Number; unit: Number of participants
Arm/Group | QGE031 | Placebo
Number analyzed (Participants) | 13 | 7
Number of participants
  Week 0 - IGA Score: 0 | 0 | 0
  Week 6 - IGA Score: 0 | 1 | 2
  Week 12 - IGA Score: 0 | 1 | 2
  Week 0 - IGA Score: 1 | 0 | 0
  Week 6 - IGA Score: 1 | 4 | 2
  Week 12 - IGA Score: 1 | 5 | 1
  Week 0 - IGA Score: 2 | 0 | 0
  Week 6 - IGA Score: 2 | 4 | 0
  Week 12 - IGA Score: 2 | 1 | 2
  Week 0 - IGA Score: 3 | 4 | 5
  Week 6 - IGA Score: 3 | 2 | 2
  Week 12 - IGA Score: 3 | 4 | 1
  Week 0 - IGA Score: 4 | 9 | 2
  Week 6 - IGA Score: 4 | 0 | 0
  Week 12- IGA Score: 4 | 0 | 0

ADVERSE EVENTS:
Groups:
- Follow-up Period: QGE031: Follow-up Period after completion of Part 1 QGE031 240 mg Q2W s.c.
- Follow-up Period: Placebo: Follow-up Period after completion of Part 1 Placebo to Match Q2W s.c.
- Follow-up Period: Open Label QGE031: Follow-up Period after completion of Part 1 Open Label QGE031 Q2W s.c.
Arm/Group | QGE031 | Placebo | Open Label QGE031 | Follow-up Period: QGE031 | Follow-up Period: Placebo | Follow-up Period: Open Label QGE031
Serious Adverse Events (participants affected / at risk) | 6/13 | 2/7 | 1/4 | 2/11 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 11/13 | 6/7 | 2/4 | 10/11 | 3/5 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 (N=13) | Placebo (N=7) | Open Label QGE031 (N=4) | Follow-up Period: QGE031 (N=11) | Follow-up Period: Placebo (N=5) | Follow-up Period: Open Label QGE031 (N=4)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 (N=13) | Placebo (N=7) | Open Label QGE031 (N=4) | Follow-up Period: QGE031 (N=11) | Follow-up Period: Placebo (N=5) | Follow-up Period: Open Label QGE031 (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Xerosis (General disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil morphology abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sciatic nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vascular dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 0 | 0
Purpura senile (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.